CLINICAL TRIAL: NCT03820453
Title: Multicentre, Randomised, Double-blind, Placebo-controlled, Parallel-group Clinical Trial to Investigate the Effectiveness of a Dietary Supplement in Increasing Libido and Sexual Function in Postmenopausal Women.
Brief Title: Clinical Trial to Investigate the Effectiveness of a Dietary Supplement in Increasing Libido and Sexual Function in Postmenopausal Women.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kern Pharma, S.L. (Industry)
Collaborators: Analysis and Research Network, S.L (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GYN-GFL-01-2018
Record Dates: First submitted 2019-01-10; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Female Sexual Arousal Disorder
MeSH Terms: interventions — Tribulus extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): One tablet per day in the morning through oral administration of a dietary supplement containing Tribulus terrestris as the main active ingredient. During three months with the possibility to extend for another three months.
  Interventions: Dietary Supplement: Tribulus Terrestris
- Control group (Placebo Comparator): One tablet per day in the morning through oral administration of Placebo. During three months.
  Interventions: Other: Placebo treatment

INTERVENTIONS:
Dietary Supplement: Tribulus Terrestris — The experimental arm will receive a dietary supplement to increase the libido and sexual function
  Arms: Active group
Other: Placebo treatment — The control arm will receive a placebo product with similar organoleptic qualities and the same posology characteristics
  Arms: Control group

SUMMARY:
This clinical Trial will assess the effects of a dietary supplement based on Tribulus terrestris on the libido and sexual function in postmenopausal women, by doing a follow up of the FSFI scale and different variables during 3 months period. Participants will be allocated to dietary supplement or placebo, and will attend to 3 visits (baseline, 6 weeks, 12 weeks and at 24 weeks optional).

ELIGIBILITY:
Inclusion Criteria:

* Women who report decreased libido and present female sexual arousal disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria
* Post-menopause.
* Age between 45 and 65 years.
* Sexually active.
* Agreement to participate and to sign the informed consent documents.

Exclusion Criteria:

* Pregnancy.
* Women who are on hormone replacement therapy or who need to start it.
* Cancer treatment or a recent history of cancer (<2 years).
* Any of the following treatments: serotonin inhibitors, GABAergics, tricyclics, antipsychotics, beta-blockers, thiazide diuretics, dopaminergics and anxiolytics for chronic problems (patients on treatment with anxiolytics without chronic problems are eligible)
* Fibromyalgia.
* Treatment for, or a history of, oestrogen-dependent cancer (breast, uterus, endometrium, etc.).
* Any comorbidity that may interfere with the pathology under study.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-08-29 (Estimated); Study Completion 2019-08-29 (Estimated)

PRIMARY OUTCOMES:
Changes of Score on the Female Sexual Function Index (FSFI) | At baseline, at 6 weeks, at 3 months and at 6 months (optional)
  Score on the Female Sexual Function Index (FSFI) Questionnaire on female libido.
  The scale has 19 questions divided in 6 Domains. Total score ranges from 2 to 36 with higher scores considered better outcome.
  Scale subdomains, their scoring range and factor to the total score is the following:
  Domain: Desire, Range [1 - 5] Factor: 0.6 Domain: Arousal, Range [0 - 5] Factor: 0.3 Domain: Lubrication, Range 0 - 5 Factor: 0.3 Domain: Orgasm Range 0 - 5 Factor: 0.4 Domain: Satisfaction Range [0 (or 1) - 5 ] Factor: 0.4 Domain: Pain Range [0-5] Factor: 0.4

SECONDARY OUTCOMES:
Variations in testosterone levels (total, bioavailable, and free) | Change from baseline to 3 months visit
  Testosterone levels (total, bioavailable and free) in blood
Change in quality of life (QoL) - Measured with Score on the Cervantes Scale. | Change from baseline, to 3 months and optional visit at 6 months
  Score on the Cervantes Scale on quality of life.
  The scale is composed of 31 questions divided in 4 domains. Each question is punctuated from 0 to 5. And total scale result ranges from 0 to 155, where 0 corresponds to the maximun QoL value and 155 worst value.
Number of adverse events | Thought the study, an average of 10 months.
  Number of adverse events (recorded in the investigator's CRF) to assess the tolerability/safety of the product
Compliance with treatment - Measured with the Morisky-Green scale | 3 months
  The Morisky-Green scale measures treatment adherence with four yes or no questions. In which yes punctuates 0 and no punctuates 1.
  Possible result values for the scale goes from 0 to 4 with 4 being a better outcome than 0.
Compliance with treatment - Recount of refounded product by patient. | 3 months
  Recount of product returned at the end of study
Compliance with treatment -Therapeutic adherence | 3 months
  Data will be collected by the investigator at participants visit with a unique question about percentage of intake. It will be considered a good compliance if 80% of the medication has been taken.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - CAP Manso, Barcelona
  - Fundació Puigvert, Barcelona
  - Hospital Clínic, Barcelona, Barcelona
  - Sexology Institute, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided